CLINICAL TRIAL: NCT06363474
Title: Cisternostomy Vs Decompressive Craniectomy for Severe Traumatic Brain Injury: Functional Outcome Comparison Using Glasgow Outcome Scale
Brief Title: Cisternostomy Vs Decompressive Craniectomy for Severe Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dr. Mustapha Shesh, Resident, M.S Neurosurgery, University of Health Sciences Lahore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHS 5532
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Severe Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Decompressive Craniectomy

STUDY DESIGN:
Intervention Model Description: The intervention model of this study is a parallel model. Patients meeting inclusion criteria are enrolled from the neurosurgery department of Punjab Institute of Neurosciences, Lahore. After obtaining consent, patients undergo detailed assessments and investigations. They're randomly assigned to Group A (decompressive craniectomy) or Group B (cisternostomy). Both procedures are performed by a single surgical team under anesthesia. Postoperatively, patients are monitored for mechanical ventilation duration, ICU and hospital stay lengths, and Glasgow Outcome Scale at discharge. This model enables outcome comparison between intervention groups while controlling confounding variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Decompressive Craniectomy (Experimental): Patients allocated to Group A will undergo decompressive craniectomy, a neurosurgical procedure involving the removal of a section of the skull (bone flap). This procedure aims to alleviate intracranial pressure (ICP) and provide additional space for the swollen brain to expand. The surgery will be performed by a single surgical team under general anesthesia. Following the procedure, patients will be closely monitored for various parameters including duration on mechanical ventilation, duration of ICU stay, duration of hospital stay, and Glasgow Outcome Scale (GOS) at the time of discharge.
  Interventions: Procedure: Decompressive Craniectomy
- Group B - Cisternostomy (Active Comparator): Arm Description: Patients allocated to Group B will undergo cisternostomy, a microsurgical technique used in neurosurgery. This procedure involves the creation of an additional space for cerebrospinal fluid (CSF) circulation to alleviate brain edema and lower intracranial pressure (ICP). The surgery will be performed by the same surgical team under general anesthesia. Postoperatively, patients will be monitored for various parameters including duration on mechanical ventilation, duration of ICU stay, duration of hospital stay, and Glasgow Outcome Scale (GOS) at the time of discharge.
  Interventions: Procedure: Cisternostomy

INTERVENTIONS:
Procedure: Decompressive Craniectomy — Patients allocated to this arm will undergo decompressive craniectomy, which involves the surgical removal of a section of the skull (bone flap). This procedure is performed to alleviate intracranial pressure (ICP) by providing additional space for the swollen brain to expand. The surgery will be performed by a single surgical team under general anesthesia. After the procedure, patients will be closely monitored for various parameters including duration on mechanical ventilation, duration of ICU stay, duration of hospital stay, and Glasgow Outcome Scale (GOS) at the time of discharge.
  Arms: Group A - Decompressive Craniectomy
Procedure: Cisternostomy — Patients allocated to this arm will undergo cisternostomy, a microsurgical technique used in neurosurgery. Cisternostomy involves the creation of an additional space for cerebrospinal fluid (CSF) circulation to alleviate brain edema and lower intracranial pressure (ICP). The surgery will be performed by the same surgical team under general anesthesia. Following the procedure, patients will be monitored for various parameters including duration on mechanical ventilation, duration of ICU stay, duration of hospital stay, and Glasgow Outcome Scale (GOS) at the time of discharge.
  Arms: Group B - Cisternostomy

SUMMARY:
The objective of this clinical study is to compare the outcomes of two neurosurgical interventions, Cisternostomy and Decompressive Craniectomy (DC), for the management of severe Traumatic Brain Injury (TBI), assessed using the Glasgow Outcome Scale (GOS). Severe TBI presents challenges in managing intracranial pressure (ICP) and cerebral perfusion, often requiring surgical intervention. DC involves the removal of a section of the skull to reduce ICP, while Cisternostomy, a technique rooted in microsurgery, aims to alleviate brain edema and lower ICP by creating additional space for cerebrospinal fluid (CSF) circulation.

This prospective study will be conducted at the Department of Neurosurgery, Punjab Institute of Neurosciences, Lahore. Patients meeting inclusion criteria will be randomized into Group A (DC) and Group B (Cisternostomy) following brain CT scans. Clinical evaluation will include regular follow-ups for 6 months post-surgery, recording data on GOS, duration of mechanical ventilation, ICU, and hospital stays. Analysis will be performed using SPSS 24, comparing outcomes between groups using Chi-square test and t-test. A significance level of p≤0.05 will be applied.

It is hypothesized that Cisternostomy, as an adjunct to traditional TBI management, will effectively reduce ICP, resulting in improved GOS and reduced complications postoperatively, including decreased duration of mechanical ventilation and ICU stay, with sustained improvement observed at 6 months

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains a major public health problem globally. Indications for neurosurgical interventions following TBI can be broadly categorised as 1) evacuation of haematoma, 2) control of traumatic intracranial pressure (ICP), 3) elevation of depressed skull, 4) repair of skull base fractures with or without dural repair, 5) treatment of hydrocephalus and 6) cranial reconstruction. Decompressive craniectomy (DC) is a neurosurgical procedure that involves the removal of a section of the skull (bone flap) and expansion duraplasty which provides additional space for the swollen brain to expand, leading to a reduction in ICP and maintained or improved cerebral perfusion pressure. As an adjunct, Cisternal opening is a well-embedded microsurgical technique in neurosurgical practice for vascular and skull base pathologies. Its application in the context of TBI, in combination with insertion of an external drain which stays in place for a few days post-operatively, has been termed cisternostomy. The objective of this study is to compare the outcome of Cisternostomy and DC for the management of severe TBI in terms of the Glasgow outcome scale (GOS). For these two groups meeting the inclusion criteria will be divided based on the lottery method after a CT scan of the brain. Group A (DC) and Group B (Cisternostomy) for severe TBI. The rationale of the procedure lies in the recognition of the important contribution of the perivascular Virchow - Robin spaces to CSF circulation. In severe TBI, increases the inter-cisternal pressure that provokes a shift of fluid from the cisternal compartment to the brain parenchyma. Although DC brings the ICP to atmospheric pressure, it does not counter react the intracerebral pressure, which causes severe brain swelling and herniation. DC may further necessitate an additional operation for cranial reconstruction, termed as cranioplasty. In this situation, cisternostomy is useful in reversing this fluid shift alleviating brain edema and thereby lowering ICP. A standard ventricular drain will be placed in the cisternal compartment which will further help in controlling the raised ICP. This study will be conducted at the Department of Neurosurgery, Punjab Institute of Neurosciences, Lahore. Clinical evaluation of the patient will be done with regular follow-up for 6 months. Data of the GOS, duration on Ventilator, ICU stay and hospital stay along with extended GOS at 6 months will be recorded and analysed. It is expected that the cisternostomy technique 3 can be considered as an adjuvant surgical strategy for severe TBI effective in reducing ICP with good GOS and a low rate of complications in the postoperative period following cisternostomy, decreased number of days on a ventilator and ICU stay with good GOS at 6 months. Performing a cisternostomy demands specific instruments and expertise in skull base and vascular surgery, making its widespread use in trauma care centers challenging. Data will be collected and analyzed by using the SPSS 24 version. Quantitative variables such as age and demographic variables will be described as Mean +/- SD for both groups. Comparison of both groups for the surgical outcome will be done by using the Chi-square test and t-test according to the nature of outcome variables. The P-value of equal or less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral mass effects such as an acute subdural haematoma greater than 10mm or a midline shift greater than 5mm on computed tomographic (CT) post-trauma.
2. Refractory ICP despite medical management (based on intracranial pressure monitoring.
3. GCS >5 and <10 following traumatic head injury
4. Age < 60 years

Exclusion Criteria:

1. Brainstem dysfunction and signs of irreversible brain damage ( i.e bilaterally non-reactive pupils)
2. Severe haemodynamic instability ( i.e polytrauma)
3. Bleeding diathesis
4. Previous head injury
5. Malignant pathology
6. Previous cranial surgery

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
comparison of patient outcomes between the two intervention groups (Decompressive Craniectomy and Cisternostomy) in terms of the Glasgow Outcome Scale (GOS). | 12 months
  The primary outcome of this study is the comparison of patient outcomes between the two intervention groups (Decompressive Craniectomy and Cisternostomy) in terms of the Glasgow Outcome Scale (GOS).

CONTACTS AND LOCATIONS:
Overall Officials: DR. MUSTAPHA SHESH, MS Neurosugery, Principal Investigator — University of Health Sciences Lahore

IPD SHARING:
Plan to Share IPD: No